CLINICAL TRIAL: NCT03968211
Title: Undetectable IgE as a Sentinel Biomarker for Humoral Immunodeficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: CSL Behring (Industry); Jeffrey Modell Foundation (Unknown)
Responsible Party: Principal Investigator, Larry Borish, MD, Professor of Medicine and Microbiology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21453
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Immune Deficiency
Keywords: immunodeficiency; IgE
MeSH Terms: conditions — Immunologic Deficiency Syndromes | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccine (Experimental): Subjects who meet enrollment criteria will be administered a single intramuscular dose of the Salmonella typhi polysaccharide vaccine
  Interventions: Biological: Salmonella typhi polysaccharide vaccine

INTERVENTIONS:
Biological: Salmonella typhi polysaccharide vaccine — Salmonella typhi polysaccharide vaccine
  Other Names: Typhim Vi

SUMMARY:
This study is trying to find out if an undetectable serum immunoglobulin E (IgE) is a biomarker, or early sign of, the development of immune deficiency.

DETAILED DESCRIPTION:
IgE is the antibody thought to be responsible for developing allergies. Undetectable serum IgE (an IgE below the lower limit of detection) is found in about 3% of the general population. In the past, it has been thought that having an undetectable IgE does not have any health impact, other than meaning that you are at low risk for having allergies. However, recent studies of patients with undetectable IgE have shown higher rates of infections, autoimmune disease and cancer.

Patients with an immune deficiency called common variable immunodeficiency (CVID) also have higher rates of infections, autoimmune disease and cancer. Recently, we have shown that most patients with CVID have a low/undetectable serum IgE.

This study is trying to find out if an undetectable serum IgE is a biomarker, or early sign of, the development of CVID or other antibody deficiencies

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Willingness and ability to comply with scheduled visits and study procedures
* Undetectable serum IgE (defined as >2 IU/mL or the lower threshold of detection)
* Normal or high serum immunoglobulins (within or above laboratory reference range for IgG, IgA, and IgM)
* patients previously seen at the University of Virginia Asthma, Allergy, and Immunology clinics where undetectable serum IgE was noted
* Control subjects must have participated in study IRB#14457 (only applicable for healthy controls in epsilon germline transcript portion of the study)

Exclusion Criteria:

* The following vulnerable populations will be excluded: pregnant women, fetuses, neonates, children, prisoners, cognitively impaired, educational or economically disadvantaged, non-English speaking subjects
* Known personal history of immunodeficiency
* Known personal history of recurrent infections
* Low serum immunoglobulins (below the laboratory reference range for IgG, IgA, or IgM)
* Recent or current treatment with systemic immunosuppression within the past 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Vaccination response | 4-6 weeks
  IgG to Salmonella typhi will be measured, with a normal response calculated as at least a 2-fold increase in IgG titers post-vaccination

SECONDARY OUTCOMES:
Epsilon germline transcript production | 3 days
  B cells isolated from subjects will be evaluated to determine their ability to produce Epsilon germline transcript in response to stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Larry Borish, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie results in a publication will be made available upon request of another researcher or if required by the publisher
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication

REFERENCES:
- [Background] Lawrence MG, Palacios-Kibler TV, Workman LJ, Schuyler AJ, Steinke JW, Payne SC, McGowan EC, Patrie J, Fuleihan RL, Sullivan KE, Lugar PL, Hernandez CL, Beakes DE, Verbsky JW, Platts-Mills TAE, Cunningham-Rundles C, Routes JM, Borish L. Low Serum IgE Is a Sensitive and Specific Marker for Common Variable Immunodeficiency (CVID). J Clin Immunol. 2018 Apr;38(3):225-233. doi: 10.1007/s10875-018-0476-0. Epub 2018 Feb 17. PMID 29453744

DOCUMENTS (1):
  • Informed Consent Form (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03968211/ICF_000.pdf